CLINICAL TRIAL: NCT00004756
Title: Randomized Study of Individualized Instruction Versus Pamphlet in Systemic Lupus Erythematosus
Brief Title: Study of Individualized Instruction Versus Pamphlet in Systemic Lupus Erythematosus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Virginia Commonwealth University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Purpose: Educational/Counseling/Training
Other Study IDs: 199/11686; VCU-92123A
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: arthritis & connective tissue diseases; disease-related problem/condition; educational needs; immunologic disorders and infectious disorders; rare disease; systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis; Connective Tissue Diseases; Immune System Diseases; Communicable Diseases; Rare Diseases

INTERVENTIONS:
Procedure: Tailored educational program
Procedure: Educational materials

SUMMARY:
OBJECTIVES:

I. Evaluate an educational program that has been pretested for cultural appropriateness and literacy requirements in patients with systemic lupus erythematosus (SLE).

II. Assess the impact of this educational program on patients with SLE, with an emphasis on recognizing cardinal symptoms, coping with fatigue, regulating medications, and communicating with the physician.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients are randomly assigned to 1 of 2 groups.

One group participates in an educational program administered and coordinated by a health educator. The program includes 1 or 2 educational sessions emphasizing practical advice, each lasting approximately 1.5 hours; social support from a patient-identified management partner; and behavioral reinforcement from health center staff, the patient partner, and written and audio materials.

The control group receives patient educational materials consistent with usual care (pamphlets).

Patients are followed at 6, 12, 24, and 36 months.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

Confirmed systemic lupus erythematosus (SLE) using American College of Rheumatology criteria

Recruitment from the Medical College of Virginia SLE registry

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 1994-12

CONTACTS AND LOCATIONS:
Overall Officials: W. Neal Roberts, Study Chair — Virginia Commonwealth University